CLINICAL TRIAL: NCT05866068
Title: Use of Clomiphene Citrate as an Inhibitor of Ovulation in an Oocyte Cryopreservation Cycle
Acronym: CCOI
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Neil Chappell (Other)
Responsible Party: Sponsor-Investigator, Neil Chappell, Physician, Woman's
Organization: Woman's (Other)
Other Study IDs: Womans
Record Dates: First submitted 2023-05-09; First posted 2023-05-19 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Infertility, Female; Infertility
MeSH Terms: conditions — Infertility, Female; Infertility | interventions — Clomiphene

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Clomiphene — Clomiphene citrate 100mg daily during IVF stimulation
  Other Names: Clomid

SUMMARY:
In vitro fertilization (IVF) has helped countless couples conceive where they otherwise were unable, but does come at a significant cost. A large portion of that cost is in the medications that allow for controlled ovarian hyperstimulation. One aspect of treatment is in ovulation inhibition to allow for supraphysiologic recruitment of oocytes prior to natural ovulation. Historically, GnRH agonist and antagonists have been used. However, these are subcutaneous injections and can be costly. Clomiphene citrate is a selective estrogen receptor modulator that acts as an estrogen antagonist in the hypothalamus and pituitary and is an inexpensive oral agent. It may be used as an inhibitor of ovulation in IVF in theory but this has never been attempted to the best of our knowledge.

DETAILED DESCRIPTION:
In vitro fertilization (IVF) has been used for over 40 years in treating infertility, and with the advent of cryopreservation, it is now possible to stimulate, retrieve and freeze oocytes for use at a later date. In fact, in late 2012 the FDA removed the experimental label from oocyte cryopreservation (OC), allowing for OC cycles to become a standard of care for patients with conditions that threaten their ovarian reserve or patients who wish to preserve their fertility electively. Currently, standard stimulation protocols for superovulation of oocytes for OC involve subcutaneous injections of GnRH agonists or antagonists to inhibit premature natural ovulation as the higher number of oocytes are recruited with gonadotropins. These medications are costly and cumbersome and therefore it is of interest to design protocols that are both easier on patient compliance and more cost effective.

Clomiphene citrate is a selective estrogen receptor modulator (SERM). It selectively binds to estrogen receptors in the hypothalamus, pituitary, ovary, endometrium, and cervix producing estrogenic and anti-estrogenic effects. However the exact mechanism of clomid is poorly understood. Multiple studies have been done through animal models. One studied showed that it inhibits the negative feedback of endogenous estrogen to subsequently increase secretion of GnRH. It is also shown to increase the frequency of GnRH, however not the amplitude [Wallach]. Current IVF protocols use either GnRH antagonist or agonist to inhibit premature ovulation. Therefore due to Clomid effect on both the hypothalamus and pituitary it could theoretically block ovulation if taken continuously to down regulate the GnRH receptors.

A study published in 1982 by Marut and Hodgen looked at the effect of high doses clomiphene in primates with normal cycles. Using high dose clomiphene (25mg daily) for five days then evaluated gonadotropins, estrogen, progesterone and preformed serial laparoscopies. In all 18 of the treatment cycles there was a delay in ovulation. Upon literature review, no other studies had been conducted looking using clomiphene citrate as a medication to inhibit ovulation during an ovarian stimulation cycle.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 18-42 years old, inclusive
* Planning to undergo IVF with egg retrieval for oocyte cryopreservation

Exclusion Criteria:

* Tobacco or illicit drug use
* History of infertility
* Prior failed IVF or OC cycle
* Drug allergy to Clomid
* Hypertension
* Migraine with aura

Ages: 18 Years to 42 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — Must be females undergoing IVF for oocyte cryopreservation
Study Population: Patients who are interested in elective oocyte cryopreservation as a pilot group to investigate the feasibility of using clomiphene as an ovulation inhibitor.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Ovulation | 3 weeks
  Evidence of premature ovulation during IVF stimulation

SECONDARY OUTCOMES:
Oocyte yield | 3 weeks
  Number of oocytes from IVF cycle
Maturity Rate | 3 weeks
  % of eggs mature / # of oocytes collected
Side effects | 3 weeks
  Number of patients reporting side effects of medication

CONTACTS AND LOCATIONS:
Locations (1):
- Womans Hospital, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No